CLINICAL TRIAL: NCT02220790
Title: Fungal Biomarkers for Diagnosis and Response to Therapy for Pediatric
Brief Title: BIOPIC: Fungal Biomarkers for Diagnosis and Response to Therapy for Pediatric Candidemia
Acronym: BIOPIC
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00056090
Record Dates: First submitted 2014-08-15; First posted 2014-08-20 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2020-08

CONDITIONS: Invasive Candidiasis
Keywords: IPFN; Pediatric; Fungal; Biomarker Assays; Candida; Pediatric ICU patient
MeSH Terms: conditions — Candidiasis, Invasive; Torulopsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to 1) define the operating characteristics of fungal biomarker assays in pediatric patients at high-risk for developing invasive candidiasis, 2) determine the change in fungal biomarker assay results in children who develop invasive candidiasis, and 3) create a biobank of blood samples from pediatric patients at high-risk for invasive candidiasis and those with invasive candidiasis for future testing of fungal biomarker assays and development of new fungal biomarker assays. The study will assemble a prospective cohort of pediatric patients at high-risk for developing invasive candidiasis. Blood samples for biomarker testing will be obtained at the time a patient has a clinical indication for blood culture attainment. Additional blood sampling will be performed on the sub-set of patients that are found to have invasive candidiasis. The sensitivity, specificity, PPV, and NPV of biomarker assays will be determined for each biomarker assay. No PHI will be stored in the database and limits on blood draws (3 ml/kg in an 8 week period) will be adhered to.

DETAILED DESCRIPTION:
This study will create an international multi-center cohort of children with new clinical concern for infection while in the hospital. Sites used are part of the International Pediatric Fungal Network (ipfn.org). The study plans to prospectively enroll pediatric patients at high-risk of developing invasive candidiasis over a four year period. The study duration per subject will be up to 14 days for blood collection and 30 days for data collection from the medical record.

For the first aim, this study will assemble a prospective cohort of pediatric patients at high-risk for developing invasive candidiasis. Blood samples for biomarker testing will be obtained within 24-hours of a patient having a clinical indication for blood culture attainment. To accomplish the second aim, additional blood sampling will be performed in the sub-set of patients that are found to have invasive candidiasis. For the third aim, remnant blood samples following biomarker testing from all consenting participants will be stored in a biobank. This biobank will be used to examine future, currently undeveloped, biomarker assays in an effort to further reduce the time to diagnosis of invasive candidiasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age > 120 days and <18 years
2. Have at least one of the following conditions:

   * admitted to a non-neonatal ICU with any underlying disease
   * being transferred imminently to a non-neonatal ICU with any underlying disease
   * have gastro-intestinal insufficiency (eg. chronic short-gut syndrome) and admitted to anywhere in the hospital
   * have a hematological malignancy (limited to AML, ALL, non-Hodgkin's lymphoma and myelodysplastic syndrome) and admitted to anywhere to the hospital
   * have a solid tumor malignancy and admitted to anywhere in the hospital
   * have a solid organ transplant and be admitted to anywhere in the hospital
   * have a hemopoietic stem cell or bone marrow transplant and be admitted to anywhere in the hospital
   * have aplastic anemia and be admitted to anywhere in the hospital
3. Have ≥ 1 central catheter (arterial or venous)
4. Have ≥ 1 blood culture drawn for clinical concern of infection at time of enrollment
5. Clinician initiates and/or changes any systemic antimicrobial therapy at time of enrollment
6. Parental/guardian permission (informed consent) and, if appropriate, child assent.
7. For Aim 2: Each of the above AND a positive blood culture or sterile site culture for Candida spp. that turns positive between day 0 and day +14.

Exclusion Criteria:

1. Diagnosis of an invasive fungal disease within the 30 days prior to the blood culture drawn of clinical concern of infection.
2. Previous inclusion in this study
3. Weight < 4 kg (Due to constraints of no more than 3 ml/kg of blood to be drawn over an 8 week period). Subjects that fall below 4 kg during the study period that blood draws are occurring will not have more than 0.75 ml/kg of blood drawn each time.
4. Patient receiving empiric anti-fungal therapy for prolonged neutropenia or fever that was started prior to the time of blood culture
5. If blood cultures obtained and anti-infectives are added/changed only as part of a local protocol and not dictated by clinical concern of infection

Ages: 120 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will create an international multi-center cohort of children with new clinical concern for infection while in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2015-01; Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
NPV, PPV, sensitivity, specificity, and threshold for positive result of fungal biomarker assays | 1 day
  Operating characteristics of fungal biomarker assays in pediatric patients at high-risk for developing invasive candidiasis

SECONDARY OUTCOMES:
change in fungal biomarker assay results | 14 days
  Measure the change in fungal biomarker assay results in those children who developed invasive candidiasis in order to monitor their response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: William J Steinbach, MD, Principal Investigator — Duke University; Brian T Fisher, DO, MPH, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (22):
- United States (19):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - All Children's Hospital, St. Petersburg, Florida
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy, Kansas City, Missouri
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York-Presbyterian Phyllis and David Komansky Center for Children's Health, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Texas Children's Hospital, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- 3rd Department Pediatrics Aristole University School of Medicine, Hippokration Hospital, Thessaloniki, Greece
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia
- Hospital d'Unverisitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Fisher BT, Boge CLK, Xiao R, Shuster S, Chin-Quee D, Allen J, Shaheen S, Hayden R, Suganda S, Zaoutis TE, Chang YC, Yin DE, Huppler AR, Danziger-Isakov L, Muller WJ, Roilides E, Romero J, Sue PK, Berman D, Wattier RL, Halasa N, Pong A, Maron G, Soler-Palacin P, Hutto SC, Gonzalez BE, Salvatore CM, Rajan S, Green M, Doby Knackstedt E, Hauger SB, Steinbach WJ. Multicenter Prospective Study of Biomarkers for Diagnosis of Invasive Candidiasis in Children and Adolescents. Clin Infect Dis. 2022 Aug 25;75(2):248-259. doi: 10.1093/cid/ciab928. PMID 35134165